CLINICAL TRIAL: NCT03627884
Title: Outcomes of the Use of Sodium Bicarbonate (8.4%) Solution as a Catheter Lock Solution as a Catheter Lock Solution to Prevent Hemodialysis Catheter Loss Due to Lumen Clot Formation
Brief Title: Outcomes of the Use of Sodium Bicarbonate (8.4%) Solution as a Catheter Lock Solution to Prevent Hemodialysis Catheter Loss Due to Lumen Clot Formation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Coney Island Hospital, Brooklyn, NY (Other)
Responsible Party: Principal Investigator, Adel S EL-Hennawy, Director of Nephrology, Coney Island Hospital, Brooklyn, NY
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-06-25
Record Dates: First submitted 2018-07-12; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: End Stage Renal Disease; Acute Renal Failure; Hemodialysis Catheter Infection; Hemodialysis Complication; Hemodialysis Access Failure; Hemodialysis Catheter-Associated Bacteremia
Keywords: Central Venous Catheters; End Stage Renal Disease; Hemodialysis; Catheter-related infection; Catheter loss due to clot formation; Acute Renal Failure
MeSH Terms: conditions — Kidney Failure, Chronic; Acute Kidney Injury; Catheter-Related Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Saline Catheter Lock Solution Group (Active Comparator): Patients receiving normal saline catheter locking solution
  Interventions: Drug: Normal Saline Catheter Lock Solution
- Sodium Bicarbonate Catheter Lock Solution (Active Comparator): Patients receiving sodium bicarbonate catheter locking solution
  Interventions: Drug: Sodium Bicarbonate Catheter Lock Solution

INTERVENTIONS:
Drug: Sodium Bicarbonate Catheter Lock Solution — Using Sodium Bicarbonate Catheter Lock Solution
  Arms: Sodium Bicarbonate Catheter Lock Solution
Drug: Normal Saline Catheter Lock Solution — Using Sodium Bicarbonate Catheter Lock Solution
  Arms: Normal Saline Catheter Lock Solution Group

SUMMARY:
Prospective, randomized, comparative clinical and open-label trial comparing sodium bicarbonate catheter lock solution (SBCLS) to normal saline catheter lock solution (NSCLS) use in HD patients with central venous catheters (CVC).

DETAILED DESCRIPTION:
A randomized, comparative clinical, open-label trial at Coney Island Hospital, in Brooklyn, NY. The study period was between October 1, 2016 and March 30, 2018, a total of 546 days. All patients provided written informed consent before enrollment. The trial protocol was approved by Maimonides Medical Center Investigational Review Board: Study #2015-06-25-CIH. Patients presenting over the age of 18 requiring hemodialysis via CVCs were eligible. One patient was excluded due to having a poor venous system with inadequate blood flow for appropriate HD. No other patient was excluded from the study.

A total of 451 patients undergoing HD with CVCs were included in the study. Patients had tunneled internal jugular vein (IJV) catheters, non-tunneled IJV catheters, and non-tunneled femoral vein catheters. All patients were randomly assigned based on simple sequential order into one of two groups: NSCLS (n = 226) and SBCLS (n = 225). NSCLS patients were assigned between October 1, 2016 and June 30, 2017. SBCLS patients were assigned between July 1 2017 and March 30, 2018. Recruitment ended based on the similar number of enrolled participants between groups. A primary or co-investigator enrolled the participant into the trial and assigned the participant to the intervention at the time of presentation. Both groups received heparin-free HD treatment. Before each HD treatment, catheters and connections were inspected for leaks, evidence of damage, exit-site infection and tunnel infection. Intraluminal SBCLS or NSCLS lock solution was removed before connecting the HD catheter to a dialysis machine prior to any treatment.

During each treatment, patients were monitored for complications and standard care was provided to every patient. After each treatment, blood was rinsed from dialysis lines with NS solution back to the patient. Upon the conclusion of treatment, all catheters were flushed and locked with 10 mL of NSCLS or SBCLS, respective of their groups. Approximately 2 mL of the injected solution remained locked within the catheter. Catheter exit site dressing changes occurred after each HD treatment.

For patients that had clotted catheters, thrombolytic therapy was not instituted. Risk assessment performed by our hospital's risk management department determined that the net risk of thrombolytic use in their opinion was greater than the risk of catheter replacement by our qualified operators.

CVCs used in the study varied according to the patient's needs and consisted of Mahurkar non-tunneled catheters and Palindrome tunneled catheters. All CVCs were inserted by an expert operator under strict aseptic protocol. Catheter care was performed by trained dialysis staff according to our hospital's Administrative Policy and Procedure Manual. At the end of dialysis, all catheters were flushed and locked with one of two solutions. SBCLS contained 7.5% or 8.4% SB at a pH of 7.0-8.5, and was used to lock SBCLS-group catheters. NSCLS contained 0.9% sodium chloride at a pH 4.5-7.0, and was used to lock NSCLS-group patient catheters. Both are sterile non-pyrogenic solutions.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting over the age of 18 requiring hemodialysis via CVCs were eligible.

Exclusion Criteria:

* Having a poor venous system with inadequate blood flow for appropriate HD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Lumen Clot Formation | Approximately 18 months
  Catheter Loss Due to Lumen Clot Formation
Catheter Related Infection | Approximately 18 months
  Catheter Loss Due to Catheter Related Infection
Malfunction | Approximately 18 months
  Catheter Loss Due to Malfunction
Overall Cause | Approximately 18 months
  Catheter Loss Due to All Causes

SECONDARY OUTCOMES:
Death | Approximately 18 months
  Number of deaths reported during the study period
Arrhythmia | Approximately 18 months
  Incidence of significant arrhythmia during dialysis requiring urgent intervention
Hemodynamic Instability | Approximately 18 months
  Incidence of extreme hypotension or hypertension requiring urgent intervention

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Hennawy AS, Frolova E, Romney WA. Sodium bicarbonate catheter lock solution reduces hemodialysis catheter loss due to catheter-related thrombosis and blood stream infection: an open-label clinical trial. Nephrol Dial Transplant. 2019 Oct 1;34(10):1739-1745. doi: 10.1093/ndt/gfy388. PMID 30668833

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-25): https://cdn.clinicaltrials.gov/large-docs/84/NCT03627884/Prot_SAP_000.pdf